CLINICAL TRIAL: NCT01280916
Title: Mindful Awareness in Body-Oriented Therapy for Women's Substance Abuse Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cynthia Price, Professor: School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33795; R21DA024771 (NIH)
Record Dates: First submitted 2011-01-12; First posted 2011-01-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-body intervention (Experimental): Mindful Awareness in Body-oriented Therapy
  Interventions: Behavioral: Mindful Awareness in Body-oriented Therapy
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Mindful Awareness in Body-oriented Therapy — 8 weekly sessions of 1.5 hours each delivered to women in substance use disorder treatment
  Arms: Mind-body intervention

SUMMARY:
The primary purpose of this exploratory and developmental study is to evaluate a mind-body intervention for relapse prevention for women in addiction treatment. The proposed intervention, Mindful Awareness in Body-Oriented Therapy (MABT), is a novel mind-body intervention designed to enhance embodiment and to facilitate mindfulness through the combination of massage, body awareness exercises and the acquisition of mindfulness skills. The treatment goals of MABT include reduction of avoidant coping responses, increase of emotional-regulation, and decrease of trauma symptoms through access to and acceptance (vs. avoidance) of sensory and emotional experience. These are thought to be important for relapse prevention given the positive association between stress, negative affect and relapse; and risk of relapse associated with PTSD symptoms. Mind-body interventions in relapse prevention are of increased clinical and scientific interest, particularly for the potential to overcome automatic response patterns that are associated with lapse and relapse in substance use treatment. This proposal falls within the current NIDA research portfolio focus on the development of interventions that will help people better cope with stress, negative affect, and trauma.

Specific Aims:

* Aim 1: To examine feasibility of recruitment to and retention in MABT as an adjunct to substance abuse treatment. Specifically, to describe a) study enrollment and barriers to recruitment, b) sample characteristics, c) response to randomization, d) session attendance, and e) loss to follow-up.
* Aim 2: To describe MABT acceptability to study participants and substance abuse treatment staff.
* Aim 3: To compare the effect of body-oriented therapy plus treatment-as-usual vs. treatment-as-usual only on reported days abstinent for overall substance use and primary drug use among women receiving substance abuse treatment, in order to estimate the effect size. Secondary analyses will examine for intervention effects on related outcomes including days abstinence on biochemical screens for substance use, body connection indicators, avoidant coping, stress reactivity, co-morbid psychological distress, and physical well-being.

ELIGIBILITY:
Inclusion Criteria:

* Female
* enrolled in weeks 1-3 of Residence XII inpatient program
* plans continued out-patient treatment at Residence XII
* willing to sign release to contact the Residence XII mental health therapist in the case of concern regarding participant safety and well being
* willing to forgo (non-study) body therapy between baseline and post-intervention assessment (3 months)
* willing to accept random assignment to study treatment conditions

Exclusion Criteria:

* Current domestic violence
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Percent Days Substance Use | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Price, PhD, Principal Investigator — University of Washington
Locations (1):
- Residence XII, Kirkland, Washington, United States